CLINICAL TRIAL: NCT01123473
Title: Effectiveness of First Line Treatment With Lapatinib and ECF/X in Histologically Proven Adenocarcinoma of the Stomach or the Esophagogastric Junction, Metastatic or Not Amenable to Curative Surgery According to HER2 and EGFR Status: a Randomized Phase II Trial
Brief Title: Epirubicin Hydrochloride, Cisplatin, and Fluorouracil or Capecitabine With or Without Lapatinib Ditosylate as First-Line Therapy in Treating Patients With Stomach Cancer or Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: company withdrew interest
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EORTC-40071; EU-21036; 2009-011580-36 (EudraCT Number)
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Gastric Cancer
Keywords: adenocarcinoma of the gastroesophageal junction; adenocarcinoma of the stomach; stage IIIA gastric cancer; stage IIIB gastric cancer; stage IIIC gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Cisplatin; Epirubicin; Fluorouracil; Lapatinib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lapatinib (Experimental): Chemotherapy + lapatinib
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: epirubicin hydrochloride; Drug: fluorouracil; Drug: lapatinib ditosylate
- Placebo (Placebo Comparator): Chemotherapy + placebo
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: epirubicin hydrochloride; Drug: fluorouracil

INTERVENTIONS:
Drug: capecitabine
Drug: cisplatin
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: lapatinib ditosylate
  Arms: Lapatinib

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin hydrochloride, cisplatin, fluorouracil, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving combination chemotherapy together with or without lapatinib ditosylate is more effective in treating patients with cancer of the stomach or gastroesophageal junction.

PURPOSE: This randomized phase II trial is studying how well epirubicin hydrochloride, cisplatin, and fluorouracil or capecitabine works when given together with or without lapatinib ditosylate as first-line therapy in treating patients with stomach cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the activity of first-line treatment comprising epirubicin hydrochloride, cisplatin, and fluorouracil or capecitabine with or without lapatinib ditosylate in patients with adenocarcinoma of the stomach or esophagogastric junction that is metastatic or not amenable to curative surgery according to HER2 and EGFR status.

Secondary

* To explore the activity of this regimen in patients who are HER2 negative by FISH, but HER2 positive by IHC (2+ and 3+) as well as patients who are HER2 positive or negative by FISH and negative by IHC (0 or 1+), but EGFR positive by FISH or by IHC (2+ and 3+).
* To assess the concordance of HER2 determination by FISH and IHC.

OUTLINE: This is a multicenter study. Patients are stratified according to institution and the combination of EGFR/HER2 status as determined by fluorescence in situ hybridization (FISH) and immunohistochemistry (IHC) assays (HER2 positive by FISH/HER2 positive by IHC 2/3+ vs HER2 negative by FISH/HER2 positive by IHC 2/3+ vs HER2 negative by IHC 0/1+/EGFR positive by FISH or by IHC 2/3+). Patients are randomized to 1 of 2 treatment arms.

* Arm I (experimental): Patients receive epirubicin hydrochloride IV and cisplatin IV on day 1; fluorouracil IV continuously on days 1-21 or oral capecitabine twice daily on days 1-21; and oral lapatinib ditosylate once daily on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (control): Patients receive epirubicin hydrochloride, cisplatin, and fluorouracil or capecitabine as in arm I. Patients also receive oral placebo once daily on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 8 weeks, every 3 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the stomach or the esophagogastric junction

  * Metastatic disease OR not amenable to curative surgery
* Tissue material for HER2 and EGFR assessment must be available
* Positive HER2 status by immunohistochemistry (IHC) OR positive EGFR by either fluorescence in situ hybridization (FISH) or IHC at time of randomization
* No clinical signs of CNS involvement

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* WBC > 3 x 10^9/L
* Absolute neutrophil count > 1.5 x 10^9/L
* Platelet count > 100 x 10^9/L
* Hemoglobin > 9 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 3 times ULN (≤ 5 times ULN in case of liver metastases)
* Serum creatinine ≤ 2.0 mg/dL
* Creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after completion of study therapy
* LVEF normal by MUGA scan or ECHO
* No serious cardiac illness within the past 6 months
* No previous or concurrent malignancies except for adequately treated cone-biopsied carcinoma in situ of the cervix or basal cell carcinoma of the skin
* Able to swallow and retain oral medication
* No history or evidence of interstitial pneumonitis or pulmonary fibrosis
* No uncontrolled infections or serious illnesses, malabsorption syndrome, or medical conditions including chronic alcohol abuse, hepatitis, HIV, and/or cirrhosis
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol or follow-up schedule

PRIOR CONCURRENT THERAPY:

* At least 12 months since prior neoadjuvant or adjuvant chemotherapy
* No other investigational drugs from 28 days prior to the first dose of study treatment until 30 days after the last dose of study treatment
* At least 30 days since prior and no concurrent drugs or herbal constituents known to be inducers or inhibitors of CYP3A4
* No prior palliative systemic chemotherapy
* No prior EGFR pathway-targeting therapy (e.g., antibodies or tyrosine kinase inhibitors)
* No concurrent traditional Chinese medicines
* No concurrent non-drug therapies such as radiotherapy (other than for pain relief) or surgery
* No other concurrent anticancer therapy or investigational agents
* No concurrent grapefruit or its juice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Response rate
Overall survival
Toxicity
Concordance of diagnostic tests

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Roth, Study Chair — Hopital Cantonal Universitaire de Geneve
Locations (4):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - U.Z. Gasthuisberg, Leuven
- Johannes Gutenberg Universitaetskliniken, Mainz, Germany
- I.P.O. Francisco Gentil - Centro De Lisboa, Lisbon, Portugal

REFERENCES:
- [Result] Roth A, Moehler MH, Mauer M, et al.: Lapatinib in combination with ECF/x in EGFR1 or HER2-overexpressing first-line metastatic gastric cancer (GC): A phase II randomized placebo controlled trial (EORTC 40071). [Abstract] J Clin Oncol 28 (Suppl 15): A-TPS205, 2010.